CLINICAL TRIAL: NCT01290744
Title: Effect of Additional Clofazimine on ENL Reactions in Leprosy
Brief Title: Effect of Additional Clofazimine on Erythema Nodosum Leprosum (ENL) Reactions in Leprosy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paul Saunderson (Other)
Responsible Party: Sponsor-Investigator, Paul Saunderson, Scientific Director, Leonard Wood Memorial
Organization: Leonard Wood Memorial (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LWM-2010-ENL
Record Dates: First submitted 2011-02-02; First posted 2011-02-07 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Borderline Lepromatous Leprosy; Lepromatous Leprosy
Keywords: leprosy; ENL; clofazimine
MeSH Terms: conditions — Leprosy, Lepromatous; Leprosy | interventions — Clofazimine; Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): These patients will receive placebo for 12 months after completion of MDT.
  Interventions: Drug: Placebo
- Clofazimine for 12 months after MDT (Experimental): Patients will be given clofazimine (100mg daily) for 12 months after completion of MDT.
  Interventions: Drug: Clofazimine

INTERVENTIONS:
Drug: Clofazimine — Clofazimine 100mg daily for 12 months after completion of MDT.
  Other Names: Lamprene
  Arms: Clofazimine for 12 months after MDT
Drug: Placebo — Daily for 12 months
  Other Names: Vitamin capsule
  Arms: Placebo group

SUMMARY:
This study is a double-blind, randomized controlled trial examining the effect on ENL reactions of giving an additional year of clofazimine after completion of MDT in leprosy.

DETAILED DESCRIPTION:
Clofazimine is an anti-bacterial agent used to treat leprosy; it is a normal component of WHO-recommended multi-drug therapy (MDT). It is also known to have a beneficial effect in one of the common immunological reactions that occur in leprosy, known as erythema nodosum leprosum, or ENL. When MDT was reduced in length from 24 to 12 months, evidence suggests that ENL became worse. This study is a double-blind, randomized controlled trial examining the effect of giving an additional year of clofazimine after completion of MDT. The endpoints are the incidence and severity of ENL over a period of 3 years in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 70 years of age
* MB leprosy
* Pretreatment BI of 4 or more at any site
* Consent

Exclusion Criteria:

* Presence of another serious illness
* Refusal of informed consent

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of ENL reactions | 2 years of follow-up
  The hypothesis is that additional clofazimine will reduce the incidence of ENL reactions in the two years following completion of MDT.

SECONDARY OUTCOMES:
Severity of ENL reactions | 2 years of follow-up
  The hypothesis is that additional clofazimine will reduce severity of ENL reactions, as well as incidence. Severity will be monitored by three indicators: 1. a rather crude clinical score (mild, moderate or severe), 2. the total dose of prednisolone given to treat ENL reactions, 3. the total duration of ENL symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marivic Balagon, MD, Principal Investigator — LWM
Locations (1):
- Cebu Skin Clinic, Cebu, Vesayas, Philippines